CLINICAL TRIAL: NCT05502289
Title: Clinical Evaluation of Delefilcon A and Verofilcon A Daily Disposable Toric Soft Contact Lenses Over One Week of Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CR-6493
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Ocular Physiology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL (Experimental): Eligible subjects will be randomized to the wear sequence (TEST/CONTROL) to wear the study lenses during each dispensing period (1 week) with a wash-out period (1 week) between wear periods.
  Interventions: Device: TEST LENS; Device: CONTROL LENS
- CONTROL/TEST (Experimental): Eligible subjects will be randomized to the wear sequence (CONTROL/TEST) to wear the study lenses during each dispensing period (1 week) with a wash-out period (1 week) between wear periods.
  Interventions: Device: TEST LENS; Device: CONTROL LENS

INTERVENTIONS:
Device: TEST LENS — DAILIES TOTAL1® for Astigmatism Contact Lenses (DT1fA)
Device: CONTROL LENS — PRECISION1™ for Astigmatism Contact Lenses (P1fA)

SUMMARY:
This is a bilateral-wear, dispensing, randomized, controlled, double-masked, 2-sequence × 2-period crossover study to evaluate ocular physiology following contact lens wear.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all the following criteria to be enrolled in the study.

The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e., not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 2 days per week during the past month.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. Have the spherical component of their vertex-corrected distance refraction must be between -0.875 to -4.625 DS (inclusive) in each eye.
7. Have the magnitude of the cylindrical component of their vertex-corrected distance refraction between 0.625 DC and 1.625 DC in both eyes.
8. Have the cylinder axis of their distance refraction between 165° and 15° (i.e., 180±15°, inclusive) or between 75° and 105° (i.e., 90±15°, inclusive) in each eye.
9. Have best corrected monocular distance visual acuity of 20/30 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study.

The subject must not:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have any ocular infection of any type.
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g., rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g., SynergEyes, SoftPerm) within the past 6 months.
6. Be currently wearing monovision or multifocal contact lenses.
7. Be currently wearing lenses in an extended wear modality.
8. Have a history of strabismus or amblyopia.
9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (6):
- United States (6):
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Sacco Eye Group, Vestal, New York
  - Professional Vision Care Inc. - Westerville, Westerville, Ohio
  - Optometry Group, LLC, Memphis, Tennessee
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 66 subjects were enrolled in this study. Of those enrolled, all 66 subjects were dispensed at least one study lens. Of those dispensed, 65 subjects completed the study while 1 subject was discontinued.
Groups:
- Test (DT1fA) \ Control (P1fA): Subjects randomized to this sequence received the Test (DT1fA) lens during the first period and then received the Control (P1fA) lens during the second period
- Control (P1fA) \ Test (DT1fA): Subjects randomized to this sequence received the Control (P1fA) lens during the first period and then received the Test (DT1fA) lens during the second period
Period: Period 1
Arm/Group | Test (DT1fA) \ Control (P1fA) | Control (P1fA) \ Test (DT1fA)
Started | 35 | 31
Completed | 34 | 31
Not Completed | 1 | 0
Not completed — Out Of Window | 1 | 0
Period: Period 2
Arm/Group | Test (DT1fA) \ Control (P1fA) | Control (P1fA) \ Test (DT1fA)
Started | 34 | 31
Completed | 34 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed one study lens.
Groups:
- Dispensed Subjects: All subjects dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.2 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 26
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 5
  White | 61
Region of Enrollment [Number; unit: Participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at every study visit (baseline, unscheduled visits and 1-week follow-up), however data collected at the 1-week follow-up is the primary endpoint. The data was then dichotomized into two groups. Those with grade 3 or higher and those with grade 2 or lower. The percentage of eyes with SLF with grade 3 or higher was reported for each lens type.
Time Frame: 1-Week Follow-up
Population: All subjects who were administered at least one study lens and had at least one observation recorded.
Measure: Number; unit: Percent
Units Other Than Participants: Eyes
Groups:
- Test (DT1fA): Subjects that wore the Test (DT1fA) lens in either the first or second period of the study.
- Control (P1fA): Subjects that wore the Control (P1fA) lens in either the first or second period of the study.
Arm/Group | Test (DT1fA) | Control (P1fA)
Number analyzed (Participants) | 66 | 66
Number analyzed (Eyes) | 132 | 132
Percent | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 8 weeks per subject.
Groups:
- Test (DT1fA): Subjects that wore the Test lens in either the first or second period of the study.
- Control (P1fA): Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test (DT1fA) | Control (P1fA)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/65
Other Adverse Events (participants affected / at risk) | 0/66 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT05502289/Prot_SAP_000.pdf